CLINICAL TRIAL: NCT03251157
Title: Dietary Intake, Allergy and Respiratory Diseases in European Adults From the GA2LEN Follow-up Survey
Brief Title: Dietary Intake in Adults From the GA2LEN Folow-up Survey
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Imperial College London (Other); Helsinki University Central Hospital (Other); Medical University of Lodz (Other); Karolinska Institutet (Other); University Ghent (Other); University of Wuerzburg (Other); Medical University of Silesia (Other); University of Coimbra (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Southern Denmark (Other); Uppsala University (Other); Umeå University (Other); Charite University, Berlin, Germany (Other); University of Southampton (Other); Göteborg University (Other); Jagiellonian University (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Vanessa Larsen, Assistant Professor in Human Nutrition, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: GA2LEN Nutrition Survey
Record Dates: First submitted 2017-08-12; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Asthma; Lung Function Decreased; Food Allergy; Allergic Sensitisation; Allergic Rhinitis; COPD; Atopy
Keywords: Asthma; Adults; Europe; Lung function; Allergy; Atopy; IgE; Sensitisation; Diet; Dietary patterns; Dietary antioxidants; Flavonoids; Fruits and vegetables; Food frequency questionnaire (FFQ); Fatty acids
MeSH Terms: conditions — Asthma; Respiratory Insufficiency; Food Hypersensitivity; Rhinitis, Allergic; Pulmonary Disease, Chronic Obstructive; Hypersensitivity | interventions — Food

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Participants had serum taken which was stored frozen and subsequently analysed in a central laboratory to estimate concentration of several biomarkers including hormones (e.g. leptin), markers of inflammation (cytokines CRP, Interleukin 6 (IL-6), Interleukin 8 (IL-8), Tumour Necrosis Factor alpha (TNF-α) Transforming Growth Factor beta (TGF-β) and Myeloperoxidase (MPO)), and serum levels of total and allergen-specific IgEs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dietary intake of various nutrients, foods and biocompounds — Participants answered a self-administered FFQ, in which they reported the usual frequency of intake of a list of 250 food items

SUMMARY:
The Nutrition Study of the GA2LEN Follow-Survey was designed to investigate the association between usual dietary intake and allergic and respiratory outcomes in adults across Europe. Within this framework, a food frequency questionnaire (FFQ) was designed to ascertain usual dietary intake of 250 food items, which was translated into the languages of the participant centres. Information on daily intake of foods, nutrients, and flavonoids was derived.

DETAILED DESCRIPTION:
Within the GA2LEN Follow-up Survey, the Nutrition Survey was aimed at assessing dietary intake in adults across European countries and its association with various outcomes of allergy and respiratory health. In absence of an internationally comparable dietary questionnaire to ascertain usual dietary intake, a single and standardized food frequency questionnaire (FFQ) was design to be used as a common instrument in all participant countries. The FFQ is comprised of 32 food sections and 250 food items. The FFQ sections were designed following the recommendations by the EFCOSUM Group, which facilitate international comparisons of dietary intake. It also included several staple foods to capture locally representative dietary intake.

Participants reported how often they had consumed each of the foods over the previous month, using eight predefined options (rarely or never, 1-3 times per month, once, 2-4, or 5-6 times per week, once, 2-3 times per day). Standard food portion sizes were used to quantify the intake following the recommendations from the UK's Food Standards Agency. Daily intake of foods (g) were estimated and macro- and micronutrient and flavonoid intakes were derived. The GA2LEN FFQ was validated in five EU countries, namely Finland, UK, Portugal, Germany, Poland, and Greece, and demonstrated to be a good tool to assess mid-term intake of foods, specifically essential polyunsaturated fatty acids (PUFAs). The instrument has also been demonstrated to be an accurate tool to assess dietary sources of flavonoids.

Various approaches were planned to derive dietary exposures and to examine their association with respiratory and allergic outcomes. These included the use of dietary patterns derived from Principal Component Analysis (PCA), a dietary inflammatory index (DII), as well as single antioxidants, and individual food items.

ELIGIBILITY:
Inclusion Criteria:

Participants aged 15-75 years old, who had responded to the GA2LEN Baseline survey and who met the definition of cases or controls (as described below)

Exclusion Criteria:

Participants who did not answer the baseline survey

Ages: 15 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The GA2LEN follow-up study was a multi-center case-control study with participants selected from the respondents to an initial cross-sectional survey of a general population of adults aged 15-74 years living in 17 European cities and completed between June 2007 and May 2009. A random sample of eligible participants who indicated a willingness to be re-contacted was selected based on their responses to the initial postal survey. The cases were participants who either had asthma, sinusitis or both and the controls (who lived in the same areas) were those who reported having neither. Each center recruited up to 120 cases each of patients with asthma only, CRS only, controls and 40 patients with both asthma and CRS based on the responses to the initial cross-sectional survey.
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Asthma score | Last 12 months
  Five questions on symptoms in the last 12 months (breathless when wheezing, woken with tightness in chest, shortness of breath while at rest, shortness of breath after exercise, woken by shortness of breath) were used to construct an asthma symptom score on a five-point scale
Chronic rhinosinusitis (CRS) | Last 12 weeks
  defined following the EP3OS criteria, that is, the presence of at least two of the following symptoms for at least 12 weeks in the past year: (i) nasal blockage, (ii) nasal discharge, (iii) facial pain or pressure or (iv) reduction in sense of smell with at least one of the symptoms being nasal blockage or nasal discharge
Lung function | Day
  Spirometric lung function (Forced Expiratory Volume in one second (FEV1), and Forced Vital Capacity (FVC)) were measured pre- and post- administration of bronchodilator (salbutamol 200 mg). Spirometric restriction was defined by an FVC below the limit of normal, chronic obstruction by an FEV1/FVC below the limit of normal. All spirometries were checked centrally for quality. Only spirometry that met the ERS/ATS criteria was accepted
Atopy | 1 day
  Skin prick tests (SPTs) to grass pollen, grass mix, Dermatophagoides pteronyssinus, Dermatophagoides farinae, cockroach (Blatella), olive, Alternaria, dog, Artemisia, birch, cat and Parietaria were conducted. A SPT was regarded as positive where the allergen weal was >1 mm more than the diluent control. Atopy was defined as any positive response to any of the allergens tested
Allergic rhinitis | Last month
  Defined based on a positive answer to the question 'Do you have any nasal allergies or hay fever'?

OTHER OUTCOMES:
Asthma | Last 12 months
  Asthma was defined as a history of ever having asthma and reporting at least one of the following symptoms in the last 12 months: wheeze or whistling in the chest, waking with chest tightness, waking with shortness of breath, and waking with an attack of coughing
IgE sensitisation | 1 day
  Serum concentrations of total IgE (geometric mean) were estimated

CONTACTS AND LOCATIONS:
Overall Officials: Peter GJ Burney, MD PhD, Study Chair — Imperial College London
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Queries on IPD from the GA2LEN Nutrition Survey may be sent to the study Principal Investigator Dr Vanessa Garcia Larsen (vgla@jhu.edu) or to the study Chair Professor Peter GJ Burney (p.burney@imperial.ac.uk)

REFERENCES:
- [Background] Bousquet J, Burney PG, Zuberbier T, Cauwenberge PV, Akdis CA, Bindslev-Jensen C, Bonini S, Fokkens WJ, Kauffmann F, Kowalski ML, Lodrup-Carlsen K, Mullol J, Nizankowska-Mogilnicka E, Papadopoulos N, Toskala E, Wickman M, Anto J, Auvergne N, Bachert C, Bousquet PJ, Brunekreef B, Canonica GW, Carlsen KH, Gjomarkaj M, Haahtela T, Howarth P, Lenzen G, Lotvall J, Radon K, Ring J, Salapatas M, Schunemann HJ, Szczecklik A, Todo-Bom A, Valovirta E, von Mutius E, Zock JP. GA2LEN (Global Allergy and Asthma European Network) addresses the allergy and asthma 'epidemic'. Allergy. 2009 Jul;64(7):969-77. doi: 10.1111/j.1398-9995.2009.02059.x. Epub 2009 Apr 7. PMID 19392994
- [Background] Garcia-Larsen V, Arthur R, Potts JF, Howarth PH, Ahlstrom M, Haahtela T, Loureiro C, Bom AT, Brozek G, Makowska J, Kowalski ML, Thilsing T, Keil T, Matricardi PM, Toren K, van Zele T, Bachert C, Rymarczyk B, Janson C, Forsberg B, Nizankowska-Mogilnicka E, Burney PGJ. Is fruit and vegetable intake associated with asthma or chronic rhino-sinusitis in European adults? Results from the Global Allergy and Asthma Network of Excellence (GA2LEN) Survey. Clin Transl Allergy. 2017 Jan 27;7:3. doi: 10.1186/s13601-016-0140-9. eCollection 2017. PMID 28149501
- [Background] Garcia-Larsen V, Luczynska M, Kowalski ML, Voutilainen H, Ahlstrom M, Haahtela T, Toskala E, Bockelbrink A, Lee HH, Vassilopoulou E, Papadopoulos NG, Ramalho R, Moreira A, Delgado L, Castel-Branco MG, Calder PC, Childs CE, Bakolis I, Hooper R, Burney PG; GA2LEN-WP 1.2 'Epidemiological and Clinical Studies'. Use of a common food frequency questionnaire (FFQ) to assess dietary patterns and their relation to allergy and asthma in Europe: pilot study of the GA2LEN FFQ. Eur J Clin Nutr. 2011 Jun;65(6):750-6. doi: 10.1038/ejcn.2011.15. Epub 2011 Mar 23. PMID 21427744